CLINICAL TRIAL: NCT06516588
Title: Post-Stroke Cognitive Impairment: Neurovascular Mechanisms and Non-Invasive Brain Stimulation
Brief Title: tDCS for Post-Stroke Cognitive Impairment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17265
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Mild Cognitive Impairment
Keywords: Post-Stroke cognitive impairment
MeSH Terms: conditions — Stroke; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- sham tDCS (Sham Comparator): Participants will receive sham (placebo) tDCS for 20 minutes, for 10 sessions
  Interventions: Device: Transcranial Dirrect Current Stimulation
- active tDCS (Experimental): Participants will receive active tDCS for 20 minutes, for 10 sessions
  Interventions: Device: Transcranial Dirrect Current Stimulation

INTERVENTIONS:
Device: Transcranial Dirrect Current Stimulation — tDCS will deliver direct current through rubber electrodes in saline-soaked sponges. Device sends a low-level current from the positive electrode, the anode, to the negative electrode, the cathode. Direct current will be transferred by a saline-soaked pair of surface sponge electrodes (35cm2) and delivered by a specially developed, battery-driven, constant current stimulator with a maximum output of 10mA. The anode will be placed over the LDLPFC and the cathode over the contralateral supra-orbital area.
  Other Names: tDCS

SUMMARY:
This study will evaluate the effects of a form of non-invasive brain stimulation on brain functioning and memory in participants with post-stroke cognitive impairment (PSCI).

DETAILED DESCRIPTION:
The goal of this study is to learn important information about the effects of electrical stimulation (Transcranial direct current stimulation (tDCS) on brain functioning in those with post-stroke cognitive impairment (PSCI). The findings will help determine how stimulation affects the brain's activity, cerebral blood flow, and circulating blood biomarkers of neuroinflammation after stroke. The study will use different forms of non-invasive brain imaging to see whether stimulation changes how the brain responds during a memory task. Functional near-infrared spectroscopy (fNIRS) and electroencephalograph (EEG) will be used, we will also collect blood samples for the biomarkers of inflammation. The study also uses cognitive tests and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1) ischemic stroke participants in sub-acute phase (at least 10 days after stroke event or discharge and under 5 months post-event) with cognitive dysfunction (MoCA <26);

Exclusion Criteria:

1. clinically significant or unstable medical or psychiatric condition;
2. diagnosis of severe depression;
3. history of relevant neurological diagnosis (e.g., epilepsy);
4. previous neurosurgical procedure with craniectomy;
5. contraindications to tDCS (implanted brain medical devices);
6. severe visual impairment, hearing impairment, aphasia, neglect or dementia.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Changes from baseline after intervention week (two weeks), one and three months
  It is a 30-point test about several cognitive domains (visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall and orientation) and a screening tool used of MCI and dementia.
NIH Toolbox | Changes from baseline after one and three months
  NIH Toolbox tests is a computarize test that acess fluid abilities (i.e., working memory, processing speed, episodic memory, and two aspects of executive functioning) and crystallized abilities (i.e., dependent upon past learning and experience), resulting in Standard Scores for these superordinate categories, as well as a total Composite score of all tests.These norms were previously reported to align with the age-corrected normative data for the traditional neuropsychological measures.

SECONDARY OUTCOMES:
Neurovascular Coupling - Cerebral blood flow (fNIRS) | Changes on fNIRS signal from baseline after after intervention week (two weeks), one and three months
  fNIRS signal will be recorded using the 16-source/16-detector system (NIRSport, NIRx)
Brain Function (EEG) | Changes on EEG signal from baseline after after intervention week (two weeks), one and three months
  EEG signal will be recorded at 1 kHz using a 16-channel system (HIAMP,g.tec).
Neurovascular Coupling - (DVA) | Changes on maximal arteriolar dilation and mean maximal venular dilation from baseline after intervention week (two weeks), one and three months
  DVA signal ill be recorded as the mean maximal arteriolar dilation and mean maximal venular dilation in response to flicker light stimulation.
Blood markers | Changes on blood marker levels from baseline after intervention week (two weeks), one and three months
  Bblood draw via venipuncture and collect up to 40mL of blood for each visit. We will separate set of plasma (for study 4), serum samples, whole blood, and blood cells (including white blood cells) , a set of each will be stored for future analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes